CLINICAL TRIAL: NCT02196584
Title: Clinical Evaluation of the Rapid Access Vitreal Injection Guide (RAVI-Guide)
Brief Title: Clinical Evaluation of the RAVI-Guide
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Dennis Han, Professor of Ophthalmology, Medical College of Wisconsin
Other Study IDs: PRO00021075
Record Dates: First submitted 2014-07-19; First posted 2014-07-22 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Retinal Diseases
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesis: The RAVI-Guide provides superior patient acceptability to the conventional lid speculum during intravitreal injections

Aims: To compare patient acceptance and procedural complication rates of the RAVI-Guide with those of the conventional lid speculum and caliper approach

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 years or older who undergo intravitreal injection for clinical indications.

Exclusion Criteria:

* Patients under the age of 18 years
* Patients unable to give informed consent
* Disorders that preclude the ability to judge pain or discomfort associated with intravitreal injection
* Disorders that preclude the ability to assess for complications of intravitreal injection
* Inability to assess the landmarks by which localization of intravitreal injection sites is determined, such as obscured corneal limbus
* Inability to communicate directly to the physician and immediately after the procedure the level of pain or discomfort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older who undergo intravitreal injection
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2014-08; Primary Completion 2015-09 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Pain severity associated with instrument type used for holding eyelids open during intravitreal injection | Within 15 minutes of injection procedure
  A pain severity scale of 0 to 10, with 0 being no pain, and 10 being worst imaginable pain, will be used to grade pain severity.

SECONDARY OUTCOMES:
Procedural complications associated with instrument use during intravitreal injection procedure | Within 15 minutes of injection procedure
  A questionnaire that queries about procedural complications will be completed by the treating physician.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis P Han, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert and Medical College of Wisconsin Eye Institute, Milwaukee, Wisconsin, United States